CLINICAL TRIAL: NCT06845943
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HCR-188 in Overweight or Obese Volunteers
Brief Title: A First-in-human Study of HCR-188 in Overweight or Obese Otherwise Healthy Volunteers Without Type 2 Diabetes
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Helicore Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCR-188-101
Record Dates: First submitted 2025-02-03; First posted 2025-02-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HCR-188 (Experimental): Single ascending dose (SAD) or multiple ascending dose (MAD) cohorts
  Interventions: Drug: HCR-188
- Placebo (Placebo Comparator): Single ascending dose (SAD) or multiple ascending dose (MAD) cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HCR-188 — Single (SAD cohorts) or multiple (MAD cohorts) subcutaneous injections
  Arms: HCR-188
Drug: Placebo — Single (SAD cohorts) or multiple (MAD cohorts) subcutaneous injections
  Arms: Placebo

SUMMARY:
This is a first-in-human study evaluating the safety, tolerability, pharmacokinetics, immunogenicity and pharmacodynamics of single and multiple doses of HCR-188 administered as subcutaneous injection(s).

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study in overweight or obese volunteers without type 2 diabetes mellitus. Up to 5 SAD cohorts and up to 5 MAD cohorts may be enrolled.

Multiple dosing regimens are planned to be evaluated in the MAD portion of the study.

The duration of the study will be approximately 20 weeks per each participant completing the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 27 to 40 kg/m2, inclusive
* Except for overweight or obese, otherwise healthy as determined by the Investigator
* Stable body weight, defined as a < 5 kg change during the 8 weeks prior to screening
* Females of childbearing potential must agree to use highly effective methods of contraception during the participation in the study
* Males must be surgically sterile, abstinent, or must agree to use highly effective methods of contraception during participation in the study

Exclusion Criteria:

* History of or active cardiovascular (CV) disease
* History of active pulmonary diseases
* History of immunosuppressive, chemotherapeutic, or radiation treatment within the last 12 months prior to Screening
* History of malignancy in the past 12 months or active malignancy
* History of bariatric surgery or use of gastric balloons
* History of diabetes mellitus Type 1 or 2
* History of chronic liver disease
* Pregnant or breastfeeding, or a positive pregnancy test at Screening
* Treatment with medications that may cause significant weight gain or weight loss

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | From the first dose and for up to 20 weeks
  Percentage of participants with treatment-emergent adverse events
Treatment-emergent adverse events resulting in treatment discontinuation | From the first dose and for up to 20 weeks
  Percentage of participants with treatment-emergent adverse events resulting in treatment discontinuation
Clinically significant laboratory values | From the first dose and for up to 20 weeks
  Percentage of participants with clinically significant laboratory values, as assessed by laboratory-based adverse events
Clinically significant vital signs | From the first dose and for up to 20 weeks
  Percentage of participants with clinically significant vital signs (blood pressure, heart rate, respiratory rate, temperature), as assessed by vital signs-related adverse events
QT interval on ECG | From the first dose and for up to 20 weeks
  Percentage of participants with an increase from baseline in the QTcF by > 60 milliseconds

CONTACTS AND LOCATIONS:
Locations (1):
- Investigative Site, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's website — https://www.helicore.com